CLINICAL TRIAL: NCT03748420
Title: A Team-Based and Technology-Driven Adherence Intervention to Improve Chronic Disease Outcomes
Brief Title: Medication Adherence Clinical Decision Support
Acronym: ADH-Wizard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A16-691; 1R01HL136937-01A1 (NIH)
Record Dates: First submitted 2018-11-14; First posted 2018-11-20 (Actual); Results first posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2023-08

CONDITIONS: Hyperlipidemia; Hypertension; Diabetes; Medication Nonadherence
Keywords: Decision Support Systems, Clinical; Cardiovascular Diseases; Cardiovascular Risk Factor; Medication Non-adherence
MeSH Terms: conditions — Hyperlipidemias; Hypertension; Diabetes Mellitus; Medication Adherence; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients in the usual care arm receive the basic cardiovascular related clinical decision support which is considered standard of care at the organization.
- Adherence Intervention (Experimental): Patients in the medication adherence enhanced clinical decision support received the enhanced decision support intervention over a 6 month period. Patients were accrued over 6 months and followed for 12 months at which point they were assessed for improved medication adherence and clinical outcomes.
  Interventions: Other: Adherence Intervention

INTERVENTIONS:
Other: Adherence Intervention — The adherence enhanced intervention consists of clinical decision support related to cardiovascular risk factors enhanced with external medication adherence information and is delivered at the point of care to the healthcare provider and patient.
  Arms: Adherence Intervention

SUMMARY:
More than 50% of adults treated for diabetes, hypertension, or lipid disorders have suboptimal medication adherence, a prominent barrier to continued improvement in chronic disease care in the United States. Primary care providers (PCPs) often fail to identify medication nonadherence and/or have insufficient time and training to address underlying reasons for it. In this project, we propose a patient-centered and technology-driven strategy to identify patients with adherence issues and apply a team approach to help them achieve evidence-based personalized goals for glucose, blood pressure, or lipids. This intervention extends the use of a widely available clinical decision support (CDS) infrastructure to support a model of care that, for the first time outside of a fully integrated care environment, will integrate pharmacists within the primary care team. The intervention relies on a continuous health informatics loop to do the following: (a) identify high-risk patients with adherence problems at the point of care by expanding the capability of an electronic medical record (EMR)-linked CDS to identify poor adherence to medications; (b) establish and maintain an auto-populating up-to-date registry of patients identified for proactive pharmacist outreach; (c) implement a pharmacist outreach strategy based on an information-motivation-behavioral (IMB) framework recommended by the World Health Organization (WHO) with demonstrated ability to influence adherence across a variety of clinical applications; and (d) coordinate care and adherence information by incorporating pharmacist assessment and action plans into CDS at subsequent office encounters.

DETAILED DESCRIPTION:
Patients are randomly allocated 1:1 through a computer-generated program to either control or intervention.

Control: All control patients will continue to receive the basic Electronic Medical Record (EMR)-linked Clinical Decision Support (CDS) tool for cardiovascular (CV) risk factor management. This CDS includes algorithmically derived identification of high CV risk patients and prioritized treatment suggestions for lipids, Blood Pressure (BP), glycemic control, weight, tobacco, and aspirin use based on distance from goal, current medications, labs, allergies, and safety considerations. The basic CDS does not include any information on medication adherence. Patients will receive basic CDS plus usual care.

Intervention: For intervention patients, the basic CDS system for CV risk-factor control is enhanced to support a team-based care model that identifies risk of non-adherence, computes adherence information and incorporates it in the CDS, creates a registry to direct proactive pharmacist outreach, and coordinates action plans. To do this, the CDS Web service will combine EMR-identified medications with Epic Medication Adherence score (e-PDC) data. Algorithms will identify poor adherence using e-PDC scores available within the Epic EMR at patient encounters. When medication adherence issues are identified, alert messages will appear on the CDS tools for patients and providers. Patients with index visits will be followed-up for 6 months as they continue to receive CDS at subsequent encounters. At 6 months, patient e-PDC as well as clinical outcomes will be reevaluated. Patients with persistent adherence issues identified are added to a registry that is used by the pharmacists to conduct outreach. Pharmacist outreach will be conducted primarily by phone, but in-person arrangements are also an option. Pharmacists conducting outreach will identify themselves to patients as part of the care team working with the primary care provider (PCP). Examples of specific action plans that may be recommended includes education, recommending lower cost alternative medications or combination medications, addressing side effects, using pill boxes, modifying pill-taking schedules and/or using reminder systems, or referrals to medication therapy management (MTM) services or health educators. Pharmacists will be guided by a script template for the phone outreach that walks them through the IMB intervention and data collection. The pharmacists involved will have full read/write access to the EMR in full compliance with HIPAA regulations. They can make medication changes through established care protocols and/or communicate with the prescriber through secure messaging or phone consultation. The date of the pharmacist outreach and actions that result from the IMB intervention will be documented in the EMR and incorporated into subsequent CDS tools and registries to reflect the new patient state.

ELIGIBILITY:
Inclusion Criteria:

* One or more of the following clinical criteria:

A. In the 12 months prior to the index visit, most recent hemoglobin A1C ≥8% AND have one or more active non-insulin glycemic medications on their electronic health record (EHR) medication list AND a potential adherence issue for one or more of these medications based on the Epic Medication Adherence score (e-PDC <80%, moderate or high confidence).

B. Two consecutive encounters with BP values ≥140/90 mm Hg AND one or more BP medications on their EHR medication list AND a potential adherence issue identified (e-PDC <80%, moderate/high confidence).

C. Meet the American College of Cardiology/American Heart Association (ACC/AHA) criteria listed below for moderate or high-intensity statin use AND a statin medication on their EHR medication list AND a potential statin adherence issue identified (e-PDC <80%, moderate/high confidence):

1. Age >21 with atherosclerotic cardiovascular disease (ASCVD) identified by a cardiovascular disease (CVD) diagnosis on the problem list or two or more International Classification of Diseases (ICD)-10 diagnostic codes in the last 2 years
2. Age >21 and LDL >190 mg/dL
3. Aged 40 to 75 AND diabetes identified by the diagnosis on the problem list or two or more ICD-10 diagnostic codes in the last 2 years
4. Aged 40 to 75 with 10-year CV Risk Score >7.5% based on the ACC/AHA 10-year ASCVD risk equation.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from the study analysis:

1. Patients enrolled in hospice,
2. Patients with active cancer or undergoing chemotherapy
3. Patients with pregnancy in the last year
4. Patients without HealthPartners insurance coverage for at least 11 of the 12 months before the index visit will be excluded from cost analysis.
5. For Statin cohort, ≥1 LDL result <100 mg/dl within 2 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5421 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J O'Connor, MD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Care System, Bloomington, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Connor PJ, Haapala JL, Dehmer SP, Chumba LN, Ekstrom HL, Asche SE, Rehrauer DJ, Pankonin MA, Pawloski PA, Raebel M, Sperl-Hillen JM. Clinical Decision Support and Cardiometabolic Medication Adherence: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jan 2;8(1):e2453745. doi: 10.1001/jamanetworkopen.2024.53745. PMID 39786775
- [Derived] Sperl-Hillen JM, Haapala JL, Dehmer SP, Chumba LN, Ekstrom HL, Truitt AR, Asche SE, Werner AM, Rehrauer DJ, Pankonin MA, Pawloski PA, O'Connor PJ. Protocol of a patient randomized clinical trial to improve medication adherence in primary care. Contemp Clin Trials. 2024 Jan;136:107385. doi: 10.1016/j.cct.2023.107385. Epub 2023 Nov 11. PMID 37956792

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were identified as eligible using an automated algorithm designed to display the adherence enhanced decision support at the point of care at a primary care clinic visit. The first visit where a participant met eligibility criteria (and prior to applying exclusion criteria) was considered their index visit. There was no direct contact between study participants and the study team. The study was granted a waiver of informed consent from HealthPartners IRB.
Pre-assignment Details: Patients were randomly allocated 1:1 through a computer generated program to either control or intervention. The number "Completed" reflects the number of participants included in the final analysis after exclusions were applied.
Groups:
- Usual Care: Patients in the usual care arm received the basic clinical decision support that is considered the standard of care at HealthPartners. Patients in this study group were accrued over 6 months and followed for 12 months at which point they were assessed for improved medication adherence and clinical outcomes.
Period: Overall Study
Arm/Group | Usual Care | Adherence Intervention
Started | 2676 | 2745
Completed | 2421 | 2486
Not Completed | 255 | 259
Not completed — No 12 month medication adherence data available | 0 | 1
Not completed — Death | 24 | 28
Not completed — Lost to Follow-up | 231 | 230

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Adherence Intervention | Total
Number analyzed (Participants) | 2676 | 2745 | 5421
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (10.6) | 57.2 (10.9) | 57.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1196 | 1235 | 2431
  Male | 1480 | 1510 | 2990
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 114 | 116 | 230
  Not Hispanic or Latino | 2045 | 2119 | 4164
  Unknown or Not Reported | 517 | 510 | 1027
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 16 | 26
  Asian | 207 | 189 | 396
  Native Hawaiian or Other Pacific Islander | 3 | 6 | 9
  Black or African American | 700 | 688 | 1388
  White | 1559 | 1630 | 3189
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 197 | 216 | 413
Region of Enrollment [Number; unit: participants]
  United States | 2676 | 2745 | 5421
Presence of cardiovascular disease (CVD) [Count of Participants; unit: Participants] | 323 | 353 | 676

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure Medication Adherence
Description: Number of patients who achieve a proportion of days covered (PDC) greater than or equal to 80% for at least one antihypertensive medication in each currently prescribed blood pressure medication class at 12 months following the index office visit date.
Time Frame: 12 months after an index visit
Population: Participants that were not at evidence-based goals for blood pressure (BP) and had PDC less than 80% with moderate to high confidence.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Adherence Intervention
Number analyzed (Participants) | 843 | 887
Participants | 396 | 470
Statistical Analysis 1: Comparison: Usual Care vs Adherence Intervention; Test type: Superiority; p = 0.0103, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [1.06 to 1.56], Standard Error of Mean 0.09845

2. Primary Outcome: Non-Insulin Glycemic Medication Adherence
Description: Number of patients who achieve a proportion of days covered (PDC) greater than or equal to 80% for at least one non-insulin glycemic medication in each currently prescribed glycemic medication class at 12 months following the index office visit date.
Time Frame: 12 months after an index visit
Population: Participants that were not at evidence-based goals for glucose (A1c) and had PDC less than 80% with moderate to high confidence.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Adherence Intervention
Number analyzed (Participants) | 596 | 628
Participants | 279 | 296
Statistical Analysis 1: Comparison: Usual Care vs Adherence Intervention; Test type: Superiority; p = 0.7967, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.82 to 1.30], Standard Error of Mean 0.1166

3. Primary Outcome: Statin Medication Adherence
Description: Number of patients who achieve a proportion of days covered (PDC) greater than or equal to 80% for a statin medication if currently prescribed at 12 months following the index office visit date.
Time Frame: 12 months after an index visit
Population: Participants that had PDC less than 80% with moderate to high confidence.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Adherence Intervention
Number analyzed (Participants) | 1039 | 1063
Participants | 529 | 586
Statistical Analysis 1: Comparison: Usual Care vs Adherence Intervention; Test type: Superiority; p = 0.0589, Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.99 to 1.41], Standard Error of Mean 0.08906

4. Primary Outcome: Mean Change in Systolic Blood Pressure
Description: Mean change in systolic blood pressure (SBP) from index to the last SBP value within 12 months after the index visit.
Time Frame: 12 months after an index visit
Population: Not at evidence-based clinical goals for SBP and had proportion of days covered (PDC) greater than or equal to 80%.
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Usual Care | Adherence Intervention
Number analyzed (Participants) | 723 | 772
mm Hg | -15.2 [-16.7 to -13.6] | -13.8 [-15.3 to -12.3]
Statistical Analysis 1: Comparison: Usual Care vs Adherence Intervention; Test type: Superiority; p = 0.21, Mixed Models Analysis; Mean Difference (Net) = 1.4, 95% CI 2-sided [-0.8 to 3.5], Standard Error of Mean 1.0871

5. Primary Outcome: Mean Change in A1c
Description: Mean change in A1c (glycated hemoglobin) value from the index visit to the last lab test within 12 months after the index visit.
Time Frame: 12 months after an index visit
Population: Participants that were not at evidence-based goals for hemoglobin A1c and had PDC less than 80% with moderate to high confidence.
Measure: Mean (95% Confidence Interval); unit: percentage of glycated hemoglobin
Arm/Group | Usual Care | Adherence Intervention
Number analyzed (Participants) | 567 | 589
percentage of glycated hemoglobin | -1.1 [-1.2 to -0.9] | -1.2 [-1.4 to -1.0]
Statistical Analysis 1: Comparison: Usual Care vs Adherence Intervention; Test type: Superiority; p = 0.20, Mixed Models Analysis; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.1234

6. Secondary Outcome: Clinic-based Medical Care Costs
Description: Change in annual clinic-based medical care costs, defined from the health system perspective.
Time Frame: 12 months after an index visit
Population: All enrolled participants that were not at evidence-based goals for blood pressure (BP) or glucose and had proportion of days covered (PDC) less than 80% with moderate to high confidence for blood pressure, glucose, or statin medications.
Measure: Mean (Standard Error); unit: US dollars
Arm/Group | Usual Care | Adherence Intervention
Number analyzed (Participants) | 2676 | 2745
US dollars | 1210.15 (40.59) | 1202.68 (44.13)
Statistical Analysis 1: Comparison: Usual Care vs Adherence Intervention; Test type: Superiority; p = 0.901, Mixed Models Analysis; Mean Difference (Net) = -7.47, 95% CI 2-sided [-124.99 to 110.04], Standard Error of Mean 59.96

ADVERSE EVENTS:
Time Frame: Safety monitoring started at a patients index date and continued for an average of 11.6 months after index date.
Description: The number of participants at Risk (safety analysis population) includes participants that were screened for eligibility and determined not eligible.
Arm/Group | Usual Care | Adherence Intervention
All-Cause Mortality (participants affected / at risk) | 24/2808 | 28/2879
Serious Adverse Events (participants affected / at risk) | 557/2808 | 559/2879
Other Adverse Events (participants affected / at risk) | 127/2808 | 127/2879
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=2808) | Adherence Intervention (N=2879)
Emergency Department visits post-index (General disorders) | 535 (535) | 543 (543)
Inpatient admissions post-index (General disorders) | 186 (186) | 178 (178)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=2808) | Adherence Intervention (N=2879)
Hypoglycemia (Endocrine disorders) | 16 | 26
Hypotension (Vascular disorders) | 22 | 16
Hypokalemia (Metabolism and nutrition disorders) | 67 | 52
Hyperkalemia (Metabolism and nutrition disorders) | 17 | 12
Hyponatremia (Metabolism and nutrition disorders) | 15 | 28
Rhabdomyolysis- post index (Musculoskeletal and connective tissue disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Because this study was conducted at a single, relatively high-performing medical group, generalizability of results to other care delivery systems or patient populations is uncertain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT03748420/Prot_SAP_000.pdf